CLINICAL TRIAL: NCT03400007
Title: Pre- and Postoperative Dynamic Floor MRI in Order to Evaluate the Anatomical and Functional Changes of the Different Pelvic Floor Organs, Before and After Prolapse Surgery.
Brief Title: Clinical and Dynamic Floor MRI Evaluation Before and After Prolapse Surgery
Status: Completed | Type: Observational
Sponsor: Tatiana Besse-Hammer (Other)
Responsible Party: Sponsor-Investigator, Tatiana Besse-Hammer, Head of clinic, Brugmann University Hospital
Organization: Brugmann University Hospital (Other)
Other Study IDs: CHUB-prolapse
Record Dates: First submitted 2018-01-09; First posted 2018-01-17 (Actual); Last update posted 2022-07-19 (Actual); Status verified 2022-07

CONDITIONS: Prolapse
Keywords: dynamic floor magnetic resonance imaging; colpocystodefecagraphy; prolapse surgery
MeSH Terms: conditions — Prolapse

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Prolapse surgery
  Interventions: Device: Dynamic floor magnetic resonance imaging; Device: Colpocystodefecography

INTERVENTIONS:
Device: Dynamic floor magnetic resonance imaging — Dynamic floor magnetic resonance imaging (MRI)
Device: Colpocystodefecography — Colpocystodefecography (CCD)

SUMMARY:
Pelvic organ prolapsed, associated with defecation disorders and urinary tracts symptoms are common and affect up to 25% of the population, mostly parous women. The pelvic floor must be seen as one entity, with multiple anatomical and physiological interactions between the various compartments (rectum, vagina, uterus and bladder) which are embedded in the same anatomical region. The often complex pathologies of this region should therefore be treated in a multidisciplinary setting.

Besides clinical evaluation, functional dynamic imaging of anorectal and pelvic floor disfunctions has an important role in the diagnosis and management of these disorders. Although the colpocystodefecography is still considered to be the golden standard in imaging this complex anatomical region, there is clearly a need for more precise imaging of the structural details, preferentially without any irradiation. Transperineal ultrasound is an option but the investigators have chosen to evaluate the use of dynamic magnetic resonance imaging. In contrast to colpocystodefecography, dynamic pelvic floor magnetic resonance imaging is an evolving technology and its precise role in functional imaging of the pelvic floor still remains to be determined.

Prolapse surgery is commonly performed and therefore it is important to assess the efficacy of the operations in correcting the anatomical defects and the symptoms associated without creating new, pelvic floor related symptoms. Few studies exist today allowing the assessment of the anatomical changes and symptoms after surgery, through abdominal or perineal approach.

This study will evaluate the reliability of the dynamic pelvic floor imaging, done in a sitting position, compared to colpocystodefecography, done in a sitting position. It will also compare clinical objective and subjective results related to pelvic floor abnormalities with imaging. Finally, it will evaluate the anatomical changes in correlation with the clinical results, organ position and inter-compartments relationships after surgery.

This study will allow to understand and explain some relapses and failures and could lead to an improvement of the indications for surgery and surgical techniques used.

ELIGIBILITY:
Inclusion Criteria:

All patients who will undergo internal or external rectal prolapse, enterocele or urogenital prolapse surgery in CHU Brugmann and CHU St Pierre.

Exclusion Criteria:

* MRI contra-indications
* Patients with prior pelvic floor surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who will be operated for symptomatic rectal intussusception or prolapse, enterocele and/or urogenital prolapse, though abdominal and persineal approach as well.
Sampling Method: Non-Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2021-10-26 (Actual); Study Completion 2021-10-26 (Actual)

PRIMARY OUTCOMES:
recto-anal angle -relax position | 6 months post surgery
  Measured by dynamic floor MRI in left lateral decubitus position (141°)
recto-anal angle -retain position | 6 months post surgery
  Measured by dynamic floor MRI in left lateral decubitus position (163°)
recto-anal angle -push position | 6 months post surgery
  Measured by dynamic floor MRI in left lateral decubitus position (165°)
recto-anal angle -relax position | 6 months post surgery
  Measured by dynamic floor MRI in sitting position (141°)
recto-anal angle -retain position | 6 months post surgery
  Measured by dynamic floor MRI in sitting position (125°)
recto-anal angle -push position | 6 months post surgery
  Measured by dynamic floor MRI in sitting position (143°)
Dynamic MRI: anterior compartment | 6 months post surgery
  From the bladder, discrete inferior descent of the pubococcygeal line: max 1/3 (yes/no)
Dynamic MRI: medium compartment | 6 months post surgery
  Vagina horizontalization (yes/no)

SECONDARY OUTCOMES:
Fecal Incontinence Severity Index (FISI) | 6 months post surgery
  This is a health tool that describes the severity of different types of incontinence for bowel contents.There are 4 items in the FISI scale with 6 answer choices. Points are awarded according to the gravity of the symptoms. The higher the FISI index (which ranges from 0 to 61), the higher the severity of the fecal incontinence.
Constipation scoring system (CCS) | 6 months post surgery
  Validated questionnaire. Minimum Score, 0 - Maximum Score, 30
Prolapse Quality of Life (P-QOL) questionnaire | 6 months post surgery
  Validated questionnaire covering nine domains: general health (1 item), prolapse impact (1 item), role (2 items), physical (2 items) and social limitations (3 items), personal relationships (2 items), emotions (3 items), sleep/energy (2 items), and severity measurement (4 items). The answers are categorized using a fourpoint Likert scale: "none/not at all," "slightly/a little," "moderately," and "a lot." A score is calculated for each domain ranging from 0 to 100. A higher score indicates a greater impairment of quality of life.
Sexual function questionnaire (PISQ-IR) | 6 months post surgery
  Validated questionnaire. The PISQ-12 measures three domains: behavioral-emotive (items 1 - 4), physical (items 5 - 9) and partner-related (items 10 - 12). It is a self-administered questionnaire, and responses are graded on a five-point Likert scale ranging from 0 (always) to 4 (never). Items 1 - 4 are reversely scored and a total of 48 is the maximum score. Higher scores indicate better sexual function.
Visual analogic Scale (VAS) | 6 months post surgery
  The VAS scale (EVA in French) is a straight line of 100 mn length. One end is the absence of pain, the other end represents unbearable pain. The patient places a mark between these 2 extremities according to the intensity of his pain at a given time.

CONTACTS AND LOCATIONS:
Overall Officials: Katleen Jottard, MD, Principal Investigator — CHU Brugmann
Locations (2):
- Belgium (2):
  - CHU Brugmann, Brussels
  - CHU St Pierre, Brussels

IPD SHARING:
Plan to Share IPD: No